CLINICAL TRIAL: NCT04202887
Title: The Effect of Low-Dose vs High-Dose Epidural Fentanyl on Gastric Emptying - A Prospective Double-Blinded Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-19-CW-004019-CTIL
Record Dates: First submitted 2019-07-17; First posted 2019-12-18 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Effects of; Anesthesia, Spinal and Epidural, in Pregnancy; Aspiration
Keywords: Anesthesia; Aspiration; Epidural opioids; Gastric ultrasound; Gastric emptying; Labor fasting guidelines
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: A double-blinded randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will be blinded to their group allocation. Upon request for labor epidural analgesia, the epidural will be performed by one of the anesthesiologists working in the delivery room who will receive an envelope with the woman's randomization. The investigator performing the gastric ultrasound will be blinded to the subject's randomization as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low Fentanyl (LF) (Active Comparator): fentanyl cumulative dose below 100mcg
  Interventions: Drug: Low Dose Fentanyl; Device: Gastric Ultrasonography
- High Fentanyl (HF) (Active Comparator): fentanyl cumulative dose above 100mcg
  Interventions: Drug: High Dose Fentanyl; Device: Gastric Ultrasonography

INTERVENTIONS:
Drug: Low Dose Fentanyl — 10ml bolus: bupivacaine 0.1% + 25mcg fentanyl, followed by a solution of bupivacaine 0.083% + fentanyl 1mcg/ml
  Arms: Low Fentanyl (LF)
Drug: High Dose Fentanyl — 10ml bolus: bupivacaine 0.1% + 100mcg fentanyl, followed by a solution of bupivacaine 0.083% + fentanyl 2mcg/ml
  Arms: High Fentanyl (HF)
Device: Gastric Ultrasonography — The Gastric US will be performed using a portable device with an abdominal probe by the same operator (EF) for all women. The Cross Sectional Area (CSA) of the antrum will be measured in the supine position with the head elevated 45 degrees. CSA will be calculated using the formula (AP x CC x pi)/4, where AC is the anterio-posterior diameter and CC the cranio-caudal diameter. Three consecutive measurements will be performed and the average of the three will be used as the final data. The cutoff used to define a "full stomach" will be a CSA above 381 mm2, which has been validated in previous studies on laboring woman. Gastric US will be performed immediately after verification of effective epidural analgesia (T0) and intrapartum, two hours after the first measurement (T2h), corresponding to a cumulative dose of 37-97mcg fentanyl in Group LF and 124-240mcg fentanyl in Group HF.

SUMMARY:
This study investigates the effect of epidural fentanyl on gastric emptying in non-fasted laboring women. Half the women will be randomized to receive low-dose epidural fentanyl (<100 mcg), and half will be randomized to receive high-dose epidural fentanyl (≥100 mcg). Gastric content will be measured by ultrasonography two hours after epidural placement and compared between the groups.

DETAILED DESCRIPTION:
Laboring women are known to be at increased risk of pulmonary aspiration in the event of general anesthesia, due to reduced lower esophageal sphincter pressure and delayed gastric emptying. Reduction in the rate of general anesthesia for cesarean delivery, improvements in airway management and premedication to improve gastric motility and increase gastric pH have greatly reduced the risk of aspiration in laboring women. This has raised questions regarding the need for restrictive fasting policies during labor, and more liberal food policies have become widespread in certain countries and birthing centers. In light of this, it is crucial to elucidate and limit any factors that may increase a woman's risk for aspiration.

Epidural opioids are usually added to the initial epidural bolus and the maintenance infusion, due to associated reduced local anesthetic dose requirements, while improving sensory block and decreasing motor block. However, systemic opioids are known to reduce gastric emptying. The effect of epidural fentanyl on gastric emptying has been investigated previously in various doses using the paracetamol absorption test. In several of these prior studies, epidural fentanyl administered in high doses (above the cut-off value of 100mcg) - either by bolus or infusion was associated with delayed gastric emptying, with no such effect with doses below this 100 mcg threshold. These studies were performed on fasting laboring women only. In addition, the paracetamol absorption test has been widely replaced by gastric ultrasonography to directly assess gastric contents by measuring the Cross-Sectional Area (CSA) of the antrum, and its feasibility has been demonstrated in laboring women.

The aim of our study is to assess the effect of high versus low dose epidural fentanyl on gastric emptying in non-fasted laboring women, using gastric ultrasonography.

Laboring women who consent to participate will be randomized to receive either high dose or low dose fentanyl in the epidural solution. A gastric ultrasound will be performed at the time of epidural placement (baseline) and two hours after the first measurement and will be compared between the two groups. Oral intake will be recorded as well in the 8 hours preceding epidural placement and between ultrasound measurements.

ELIGIBILITY:
Inclusion Criteria:

* Laboring women ≥18 years of age
* ≥37 weeks gestation
* Singleton pregnancy with cephalad fetus
* Cervical dilatation less than 5cm
* Request for epidural analgesia

Exclusion Criteria:

* Contraindications to neuraxial analgesia
* Chronic opioid consumption
* Increased risk of emergency cesarean delivery - Trial of labor after cesarean delivery (TOLAC), twin pregnancy, non-reassuring fetal heart rate (NRFHR), dysfunctional labor, estimated fetal weight>4000g, body mass index (BMI) ≥ 40kg/m2.
* Increased risk of aspiration - Disorders of the upper gastrointestinal tract (severe gastro-esophageal reflux, history of bariatric surgery), neurological and endocrine disorders associated with gastroparesis (such as multiple sclerosis, diabetes with autonomic neuropathy)
* BMI > 40kg/m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
CSA two hours after epidural placement | 2 hours after epidural placement
  CSA measured by ultrasonography two hours after first measurement (at T2h) in "High dose Fentanyl" (HF) versus "Low dose Fentanyl" (LF)

SECONDARY OUTCOMES:
Change in CSA from baseline in HF versus LF | Baseline and at 2 hours
  Comparison of CSA at 2h for subgroups - LF/Empty vs. HF/Empty and of LF/Full vs. HF/Full , and comparison of CSA-baseline vs. CSA-2h for each subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, M.D., Study Chair — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiszer E, Aptekman B, Baar Y, Weiniger CF. The effect of high-dose versus low-dose epidural fentanyl on gastric emptying in nonfasted parturients: A double-blinded randomised controlled trial. Eur J Anaesthesiol. 2022 Jan 1;39(1):50-57. doi: 10.1097/EJA.0000000000001514. PMID 33852498

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04202887/Prot_SAP_000.pdf